CLINICAL TRIAL: NCT03226405
Title: Patient Navigation to Improve Patient-Centered Cancer Care
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Sanja Percac-Lima, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 17-183
Record Dates: First submitted 2017-07-19; First posted 2017-07-21 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Cancer
Keywords: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Patient Navigation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient Navigation Program (Experimental): * The study team will identify, track, and provide navigation for all adult patients referred to Cancer Center from the CHC and community partners for cancer treatment.
  * The Patient Navigation Program include
    * Education,
    * Appointment reminders,
    * Help with insurance,
    * Transportation,
    * Navigating the Cancer Center,
    * Assisting in finding appropriate child care,
    * Interpreting,
    * Connecting the patient to psychosocial and/or palliative care teams,
    * Physically escorting the patient to appointments
  Interventions: Other: Patient Navigation Program
- Standard of Care (Active Comparator): * The patients will receive enhanced usual care,
  * This consist of personal phone call reminders about upcoming appointments at the MGH Cancer Center
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Patient Navigation Program — PN program improve access, timeliness and adherence with cancer treatment
  Arms: Patient Navigation Program
Other: Usual Care — the standard of care provided by the institution
  Arms: Standard of Care

SUMMARY:
The MGH Cancer Center's patient navigation (PN) program, utilizes specially trained community-based personnel to improve cancer care in underserved communities by increasing cancer screening and removing barriers to timely care. This program incorporate rigorous evaluation to demonstrate the impact of innovation in healthcare delivery.

DETAILED DESCRIPTION:
This program allow cancer patients from MGH Community Health Centers (CHC) and surrounding communities who experience barriers to accessing care, including poverty, and limited English proficiency, and provide them navigation to receive timely, guideline-concordant treatment at MGH Cancer Center. By offering these vulnerable individuals a patient-centered approach to treatment, The investigators aim to promote patient engagement and increase access throughout the continuum of cancer care.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age 18 and older)
* Newly diagnosed with cancer referred from Massachusetts General Hospital (MGH) community health centers in

  * Revere
  * Chelsea
  * Charlestown
  * surrounding communities referred to receive cancer treatment at the MGH Cancer Center

Exclusion Criteria:

-Patients that primary care providers exclude

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2020-10-02 (Estimated); Study Completion 2023-10-02 (Estimated)

PRIMARY OUTCOMES:
Adherence With Cancer Treatment | 2 years
  Adherence with cancer treatment will be measured as no-show rate to scheduled oncology appointments.
The Time From Cancer Diagnosis To First Oncology Appointment | 2 Years
  Length of time in days from cancer diagnosis to first completed oncology appointment.

SECONDARY OUTCOMES:
Health Related Quality Of Life | 2 years
  Health related quality of life measured via the validated Functional Assessment of Cancer Therapy - General (FACT-G).
Overall Survival | 2 years
  Overall survival rate of the study population.
Proportion Of Patients Enrolled In Clinical Trials | 2 years
  Proportion of participants in the study that enroll on a clinical trial.
Overall Missed Health Care Visits | 2 years
  Number of scheduled health care visits missed by enrolled patients.
Emergency Department Visits | 2 years
  Number of emergency department visits by enrolled patients.
Unplanned Hospitalizations/Readmissions | 2 years
  Number of unplanned hospitalizations and/or readmissions by enrolled patients.
Inpatient Hospitalization Length Of Stay. | 2 years
  Number of days enrolled patients spent as a hospitalized inpatient.
Patient Satisfaction With Patient Navigation Program (PNP) | 2 years
  Patient satisfaction with patient navigation program (PNP) to be measured via the validated Patient Satisfaction with Navigation - 1 (PSN-1).
Patient Engagement In Care | 2 years
  Patient engagement in care will be measured using the validated Perceived Efficacy in Patient-Physician Interactions (PEPPI) metric.
Patient's Financial Burden | 2 years
  Patient financial burden will be measured using the validated Comprehensive Score for Financial Toxicity (COST) instrument.
Patient Satisfaction with Cancer Care | 2 years
  Patient satisfaction with cancer care to be measured using the validated Cancer-Related Care Survey.

CONTACTS AND LOCATIONS:
Overall Officials: Sanja Percac-Lima, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No